CLINICAL TRIAL: NCT02707692
Title: Perturbing the HIV Reservoir With Immune Stimulation
Brief Title: Perturbing of HIV Reservoir With Immune Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, David Smith, Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 160089; 1R01AI118422-01A1 (NIH)
Record Dates: First submitted 2016-02-23; First posted 2016-03-14 (Estimated); Results first posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: AIDS; HIV
Keywords: HIV; AIDS; Immune Stimulation; HIV Reservoir
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — fluarix; Pneumococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Pneumococcal, then Influenza, then Placebo vaccination (Other): Participants first received a 0.5 mL injection of Pneumococcal vaccine (Pneumovax-23®). After a washout period of at least 6 weeks, they then received a 0.5 mL injection of Influenza vaccine (Fluarix®, GSK). After another washout period of at least 6 weeks, the participant received a 0.5 mL injection of saline (placebo).
  Interventions: Biological: Fluarix; Biological: Pneumovax; Other: Placebo
- Pneumococcal, then Placebo, then Influenza vaccination (Other): Participants first received a 0.5 mL injection of Pneumococcal vaccine (Pneumovax-23®). After a washout period of at least 6 weeks, they then received a 0.5 mL injection of saline (placebo). After another washout period of at least 6 weeks, the participant received a 0.5 mL injection of Influenza vaccine (Fluarix®, GSK).
  Interventions: Biological: Fluarix; Biological: Pneumovax; Other: Placebo
- Influenza, then Pneumococcal, then Placebo vaccination (Other): Participants first received a 0.5 mL injection of Influenza vaccine (Fluarix®, GSK). After a washout period of at least 6 weeks, they then received a 0.5 mL injection of Pneumococcal vaccine (Pneumovax-23®). After another washout period of at least 6 weeks, the participant received a 0.5 mL injection of saline (placebo).
  Interventions: Biological: Fluarix; Biological: Pneumovax; Other: Placebo
- Influenza, then Placebo, then Pneumococcal vaccination (Other): Participants first received a 0.5 mL injection of Influenza vaccine (Fluarix®, GSK). After a washout period of at least 6 weeks, they then received a 0.5 mL injection of saline (placebo). After another washout period of at least 6 weeks, the participant received a 0.5 mL injection of Pneumococcal vaccine (Pneumovax-23®).
  Interventions: Biological: Fluarix; Biological: Pneumovax; Other: Placebo
- Placebo, then Pneumococcal, then Influenza vaccination (Other): Participants first received a 0.5 mL injection of saline (placebo). After a washout period of at least 6 weeks, they then received a 0.5 mL injection of Pneumococcal vaccine (Pneumovax-23®). After another washout period of at least 6 weeks, the participant received a 0.5 mL injection of Influenza vaccine (Fluarix®, GSK).
  Interventions: Biological: Fluarix; Biological: Pneumovax; Other: Placebo
- Placebo, then Influenza, then Pneumococcal vaccination (Other): Participants first received a 0.5 mL injection of saline (placebo). After a washout period of at least 6 weeks, they then received a 0.5 mL injection of Influenza vaccine (Fluarix®, GSK). After another washout period of at least 6 weeks, the participant received a 0.5 mL injection of Pneumococcal vaccine (Pneumovax-23®).
  Interventions: Biological: Fluarix; Biological: Pneumovax; Other: Placebo

INTERVENTIONS:
Biological: Fluarix — Intramuscular injection with Fluarix® .
Biological: Pneumovax — Intramuscular injection with Pneumovax.
Other: Placebo — Intramuscular injection with sterile saline (placebo).

SUMMARY:
The purpose of this study is to determine the impact of Pneumococcus and Influenza vaccines on the HIV transcriptional activity in individuals who are virologically suppressed for at least 48 weeks on similar ART. The proposed study is a randomized double-blinded control trial conducted over 28 weeks. Randomized interventions will be injections of Influenza vaccine, Pneumococcal vaccine, and Placebo. Each participant will receive each injection but in a randomized order.

DETAILED DESCRIPTION:
Title: Perturbing the HIV Reservoir

Sample Size: 56

Study Population: HIV-infected individuals between 18 and 65 years old who started similar antiretroviral therapy (ART) during chronic infection and remained virally suppressed for at least 48 weeks before enrollment. Participants will have CD4 >250 cells/μl at enrollment and a CD4 nadir >100 cells/μl.

Participating Sites: UCSD's Antiviral Research Center (AVRC)

Study Design: The proposed study is a randomized double-blinded control trial conducted over 28 weeks. Randomized interventions will be injections of Influenza vaccine, Pneumococcal vaccine, and Placebo. Each participant will receive each injection but in a randomized order.

Schedule of Evaluations: Study evaluations will be based on three 30 day cycles (Influenza vaccine, Pneumococcus vaccine, Placebo in random order) over 28 weeks of the RCT. Pre injection: one paired blood and genital secretion sample will be collected before each injection. Post-injection: paired blood and genital secretion samples will be collected on days 2, 4, 7, 14 and 30 after each injection.

Study Duration: 240 weeks

Study Regimen/Intervention: This is a double blind RCT of two vaccines (Pneumovax®23 and Fluarix®) plus placebo (sterile saline injection). Study participants will be followed for 28 weeks after enrollment. During this 28-week period, blood and genital secretion samples will be collected on day 0 and five subsequent time points after each injection (days 2, 4, 7, 14 and 30). Injections (vaccine or placebo) will be administered 12 weeks apart and in a random order, to minimize a possible bias due to the order of the vaccines.

Primary Objective: To determine the impact of Pneumococcus and Influenza vaccines on the HIV transcriptional activity in individuals who are virologically suppressed for at least 48 weeks on similar ART.

Primary Outcome: Average level of CD4+ T cell-associated HIV RNA transcription measured at days 2, 4, 7, 14 and 30 after each injection.

ELIGIBILITY:
Inclusion Criteria

1. Documented HIV-1 infection more than 365 days ago (HIV antibody or viral load positive).
2. Capable of signing written informed consent.
3. Documented viral s suppression for at least 48 weeks (≤50 copies/mL)
4. Men and women between 18 and 65 years of age.
5. Read and comprehend English.
6. Documented CD4 count at enrollment (>250 cells/µl)
7. Reported CD4 nadir >100 cells/µl.
8. Received seasonal flu vaccination at least 6 weeks prior to first trial injection (and not more recently)
9. Received vaccination for pneumococcal disease at least 12 months prior to first trial injection (and not more recently)
10. Started ART during chronic infection (> 6 months from estimated date of injection)

Exclusion Criteria

1. Uncontrolled psychiatric condition.
2. Under the influence of drug(s) or alcohol at time of screening.
3. Any condition that, in the opinion of the investigator, would limit follow-up and adequate consent.
4. History of allergic reactions to any of the proposed vaccines or egg allergy.
5. History of Gullian Barre syndrome
6. Receiving immunosuppressive medications.
7. Pregnancy or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2022-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD Antiviral Research Center (AVRC), San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gianella S, Anderson C, Chaillon A, Wells A, Porrachia M, Caballero G, Meneses M, Lonergan J, Woodworth B, Gaitan NC, Rawlings SA, Muttera L, Harkness L, Little SJ, May S, Smith D. Impact of influenza and pneumococcal vaccines on HIV persistence and immune dynamics during suppressive antiretroviral therapy. AIDS. 2024 Jul 1;38(8):1131-1140. doi: 10.1097/QAD.0000000000003882. Epub 2024 Mar 22. PMID 38526550

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates: 2016 to 2020 Recruitment location: Conducted in HIV clinics and at clinical trial site, UC San Diego AntiViral Research Center in San Diego, CA
Pre-assignment Details: Participants had a wash out period of no less than 4 weeks between vaccination series. Participants were excluded from the study before randomization and study assignments if their HIV viral loads were detectable from blood samples collected at screening.
Period: Cycle 1 (30 Days)
Arm/Group | Pneumococcal, Then Influenza, Then Placebo Vaccination | Pneumococcal, Then Placebo, Then Influenza Vaccination | Influenza, Then Pneumococcal, Then Placebo Vaccination | Influenza, Then Placebo, Then Pneumococcal Vaccination | Placebo, Then Pneumococcal, Then Influenza Vaccination | Placebo, Then Influenza, Then Pneumococcal Vaccination
Started | 9 | 9 | 9 | 9 | 9 | 9
Completed | 8 | 6 | 8 | 9 | 8 | 8
Not Completed | 1 | 3 | 1 | 0 | 1 | 1
Period: Washout Between Cycles 1 and 2 (>=6 Wks)
Arm/Group | Pneumococcal, Then Influenza, Then Placebo Vaccination | Pneumococcal, Then Placebo, Then Influenza Vaccination | Influenza, Then Pneumococcal, Then Placebo Vaccination | Influenza, Then Placebo, Then Pneumococcal Vaccination | Placebo, Then Pneumococcal, Then Influenza Vaccination | Placebo, Then Influenza, Then Pneumococcal Vaccination
Started | 8 | 6 | 9 | 9 | 8 | 8
Completed | 7 | 6 | 9 | 8 | 7 | 8
Not Completed | 1 | 0 | 0 | 1 | 1 | 0
Period: Cycle 2 (30 Days)
Arm/Group | Pneumococcal, Then Influenza, Then Placebo Vaccination | Pneumococcal, Then Placebo, Then Influenza Vaccination | Influenza, Then Pneumococcal, Then Placebo Vaccination | Influenza, Then Placebo, Then Pneumococcal Vaccination | Placebo, Then Pneumococcal, Then Influenza Vaccination | Placebo, Then Influenza, Then Pneumococcal Vaccination
Started | 7 | 6 | 9 | 8 | 7 | 8
Completed | 6 | 6 | 9 | 7 | 4 | 7
Not Completed | 1 | 0 | 0 | 1 | 3 | 1
Period: Washout Between Cycles 2 and 3 (>=6 Wks)
Arm/Group | Pneumococcal, Then Influenza, Then Placebo Vaccination | Pneumococcal, Then Placebo, Then Influenza Vaccination | Influenza, Then Pneumococcal, Then Placebo Vaccination | Influenza, Then Placebo, Then Pneumococcal Vaccination | Placebo, Then Pneumococcal, Then Influenza Vaccination | Placebo, Then Influenza, Then Pneumococcal Vaccination
Started | 7 | 6 | 9 | 7 | 6 | 7
Completed | 7 | 6 | 9 | 5 | 6 | 6
Not Completed | 0 | 0 | 0 | 2 | 0 | 1
Period: Cycle 3 (30 Days)
Arm/Group | Pneumococcal, Then Influenza, Then Placebo Vaccination | Pneumococcal, Then Placebo, Then Influenza Vaccination | Influenza, Then Pneumococcal, Then Placebo Vaccination | Influenza, Then Placebo, Then Pneumococcal Vaccination | Placebo, Then Pneumococcal, Then Influenza Vaccination | Placebo, Then Influenza, Then Pneumococcal Vaccination
Started | 7 | 6 | 9 | 5 | 6 | 6
Completed | 5 | 5 | 9 | 5 | 5 | 5
Not Completed | 2 | 1 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pneumococcal, Then Influenza, Then Placebo Vaccination | Pneumococcal, Then Placebo, Then Influenza Vaccination | Influenza, Then Pneumococcal, Then Placebo Vaccination | Influenza, Then Placebo, Then Pneumococcal Vaccination | Placebo, Then Pneumococcal, Then Influenza Vaccination | Placebo, Then Influenza, Then Pneumococcal Vaccination | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (13.4) | 42.9 (9.5) | 42.2 (13.4) | 44.3 (10.2) | 46.9 (10.1) | 48.0 (10.9) | 45.0 (11.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 6 | 8 | 8 | 8 | 7 | 8 | 45
  Gender: Female | 3 | 1 | 0 | 0 | 1 | 1 | 6
  Gender: Trans or non-binary | 0 | 0 | 1 | 1 | 1 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 3 | 4 | 5 | 4 | 27
  Not Hispanic or Latino | 3 | 4 | 6 | 5 | 4 | 5 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 2 | 0 | 2 | 8
  White | 8 | 7 | 7 | 6 | 9 | 5 | 42
  More than one race | 0 | 0 | 0 | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants] — Recruitment occurred in San Diego, California and blood collection occurred via standard phlebotomy
  participants
    United States | 9 | 9 | 9 | 9 | 9 | 9 | 54
Virologically suppressed [Count of Participants; unit: Participants]
  Suppressed (< 50 copies/ml) | 9 | 9 | 9 | 9 | 8 | 8 | 52
  Viremic (>= 50 copies/ml) | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 1
CD4 Counts [Mean (Standard Deviation); unit: cells/microliters] — Population: The CD4 count was not ascertained for one participant in Arm 5 ("Placebo, then Pneumococcal, then Influenza vaccination").
  cells/microliters
    number analyzed (Participants) | 9 | 9 | 9 | 9 | 8 | 9 | 53
    (all) | 785.4 (248.5) | 814.9 (267.9) | 798.4 (280.0) | 724.4 (256.7) | 753.8 (242.4) | 639.9 (222.1) | 752.8 (248.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Vaccination (Day 0) in Mean CD4+ T Cell-associated HIV RNA Transcription at Day 7
Description: CD4+ T cell-associated HIV RNA was measured before vaccination on Day 0 and again on Day 7. The Day-0 measure of CD4+ T cell-associated HIV RNA transcription was subtracted from the Day-7 measure.
Time Frame: Day 0 and Day 7
Population: Within each cycle, all participants who received the vaccination and completed the Day-7 visit were included in the analysis.
Measure: Mean (Standard Deviation); unit: HIV RNA copies per million cell
Groups:
- Pneumococcal Vaccine: Participants received a 0.5 mL injection of Pneumococcal vaccine (Pneumovax-23®) and a 0.5 mL of saline (placebo) with at least 6 weeks of washout between injections, in random order.
- Influenza Vaccine: Participants received a 0.5 mL injection of Influenza vaccine (Fluarix®, GSK) and a 0.5 mL of saline (placebo) with at least 6 weeks of washout between injections, in random order.
- Placebo: Participants received a 0.5 mL injection of saline (placebo).
Arm/Group | Pneumococcal Vaccine | Influenza Vaccine | Placebo
Number analyzed (Participants) | 42 | 44 | 45
HIV RNA copies per million cell | -471.8 (2998.0) | -45.9 (243.2) | 332.3 (2266.4)
Statistical Analysis 1: Comparison: Pneumococcal Vaccine vs Placebo; Primary hypothesis: Participants will have a higher absolute difference in levels of CD4+ T cell-associated HIV RNA transcription seven days after receiving either Pneumococcal or Influenza vaccinations, when compared to seven days after receiving placebo; Test type: Superiority; p = 0.32, Paired t-test, 2 sided; Mean Difference (Final Values) = -988.0, 95% CI 2-sided [-2996.3 to 1020.3]
Statistical Analysis 2: Comparison: Influenza Vaccine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.31, Paired t-test, 2 sided; Mean Difference (Final Values) = -405.0, 95% CI 2-sided [-1199.7 to 389.7]

ADVERSE EVENTS:
Time Frame: From baseline until the end of Cycle 3 (up to 417 days on study)
Groups:
- Pneumococal Vaccine: Participants received a 0.5 mL injection of Pneumococcal vaccine (Pneumovax-23®).
- Influenza Vaccine: Participants received a 0.5 mL injection of Influenza vaccine (Fluarix®, GSK).
Arm/Group | Pneumococal Vaccine | Influenza Vaccine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45 | 0/48
Serious Adverse Events (participants affected / at risk) | 1/45 | 0/45 | 0/48
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45 | 0/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pneumococal Vaccine (N=45) | Influenza Vaccine (N=45) | Placebo (N=48)
Elevated ALT/AST (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/92/NCT02707692/Prot_SAP_000.pdf